CLINICAL TRIAL: NCT03526380
Title: Translation of Opiate Overdose Prevention Strategies
Brief Title: The OPT-IN Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amy S.B. Bohnert, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R49CE002099 (NIH)
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Opioid-Related Disorders
Keywords: Drug overdose; Substance-Related Disorders; Chemically-Induced Disorders; Risk Reduction Behavior; Harm Reduction
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Substance-Related Disorders; Chemically-Induced Disorders; Risk Reduction Behavior; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants receive the OPT-IN Brief Intervention.
  Interventions: Behavioral: Behavioral: the OPT-IN Intervention
- Control (No Intervention): Participants will only complete the baseline and follow-up surveys.

INTERVENTIONS:
Behavioral: Behavioral: the OPT-IN Intervention — A private one-on-one brief motivational interviewing intervention administered by non-research staff at community organizations. This will take up to 30 minutes to complete. The goal of the intervention is to improve opioid safety and reduce related overdoses among those who has a history of misusing opioids (prescription and illicit). The session will use techniques to change behavior in a respectful, non-confrontational, and non-judgmental manner. This intervention will also seek to empower participants by providing content on bystander response as well as peer outreach, which emphasizes ways to discuss overdose risk with others at risk for overdose.
  Arms: Treatment

SUMMARY:
Prescription opioid overdose represents a public health crisis. A number of efforts have been implemented to address opioid prescribing and opioid risk mitigation strategies for prescribers, but relatively few efforts have sought to address this problem directly with individuals who use opioids. This gap likely fails to fully address the inherent reinforcing nature of the medications that make it challenging to reduce use.

The specific aim of this study is to pilot test a toolkit that pairs an intervention with the distribution of naloxone. External facilitation (supervision check-ins) will aid translation to delivery by non-research staff. Firstly, data will be collected from participants over time as a control group, prior to training site staff. Next, non-research staff will be trained on the intervention. Staff at the site will use the online "toolkit" developed in the beginning of this project to deliver the interventions and naloxone to their clients/patients as part of usual care. After staff at the site(s) are trained, additional data will be collected from participants during the intervention period and after 3-months.

DETAILED DESCRIPTION:
Based on feedback from non-research site staff, the OPT-IN Project implementation package was tailored for optimal delivery in the site setting. The translation strategy will be evaluated using the RE-AIM framework, which includes Reach (e.g., number of individuals receiving intervention), Effectiveness (e.g., patient/client outcomes), Adoption (e.g., numbers trained), Implementation (e.g., fidelity of intervention delivery) and Maintenance (e.g., sustained in routine practice over time) with mixed qualitative and quantitative methods with intervention recipients.

ELIGIBILITY:
Inclusion Criteria:

* Speaks English Fluently
* Receiving services at one of the investigator's partner sites
* History of opioid use

Exclusion Criteria:

* Medically unstable
* Prisoners
* Inability to speak and understand English
* Inability to give informed, voluntary, written consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Overdose Risk Behaviors (ORB) | 3 months post-baseline
  The ORB measures change over time for prescription opioid use, specific to type of opioid use, combination with other substances, route, and if they use alone. This scale is a total sum of 9 items assessing participant's self-report of engaging in behavior that increases risk for overdose. Higher scores indicate greater risk for overdose. The range for this measure is 0 to 32 in one assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States